CLINICAL TRIAL: NCT02772523
Title: Control and Intervention Programme on Alzheimer's Disease Risk Factors
Acronym: ALFAlife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALFAlife/BBRC2015
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease
Keywords: Primary Prevention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other)
  Interventions: Other: Lifestyle recommendations

INTERVENTIONS:
Other: Lifestyle recommendations — Dietary, and physical, cognitive and social activity recommendations

SUMMARY:
Recent epidemiologic studies are identifying a number of modifiable risk and protective factors that may influence in the incidence of Alzheimer's disease (AD). Therefore, the combination of an early detection of individuals at risk together with interventional studies targeted to the control of modifiable risk factors makes primary prevention programmes to become a new and real therapeutic strategy.

In this scenario, the investigators have designed the ALFAlife study, a programme of control and intervention on the modifiable AD risk factors. Throughout this study, participants will be given a number of healthy lifestyle guidelines that are personalised depending on their specific risk profile. These guidelines refer to smoking and dietary habits and physical, cognitive and social activity. The investigators hypothesis is that the follow-up of these guidelines will favor a change of participants' lifestyle habits towards healthier ones. In addition, the investigators hypothesise that changes in these lifestyle habits will have an effect on objective physiological measures (such as blood pressure and cholesterol levels).

ELIGIBILITY:
Inclusion Criteria:

* Participants in the ALFA study (NCT01835717)
* Computer literacy
* Accept study's tests and procedures
* Signature of informed consent

Exclusion Criteria:

* Cognitive impairment assessed by clinical criteria that, according to the investigator's evaluation could interfere with the study's follow-up.
* Anxiety or depression assessed by clinical criteria that, according to the investigator's evaluation could interfere with the study's follow-up.
* Visual and/or hearing impairment severe enough to impede tests realization.
* Major psychiatric or neurological disorder or other diseases that according to the investigator's evaluation could interfere with the study's follow-up.
* Antecedents of infarction, ischemic heart disease, stroke, peripheral vascular disease, stent or aneurysm clip

Ages: 45 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in Short Version of the Minnesota Leisure Time Physical Activity Questionnaire | 1 year; change between baseline and one year after
Change in 14-item mediterranean diet Questionnaire | 1 year; change between baseline and one year after
Change in Lifestyle Activities Questionnaire (LAQ) | 1 year; change between baseline and one year after

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Catalonia, Spain